CLINICAL TRIAL: NCT00909636
Title: A Double-Blind, Randomized, Placebo-Controlled Study of the Safety, Tolerability, and Pharmacokinetics of Multiple Doses of ABT-333 in Healthy Adults
Brief Title: A Study to Assess the Safety, Tolerability, and Pharmacokinetics of Multiple Ascending Doses of the ABT-333 Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Daniel Cohen, MD/Study Medical Director, Abbott
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M11-031
Record Dates: First submitted 2009-05-27; First posted 2009-05-28 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-09

CONDITIONS: HCV Infection
Keywords: multiple ascending doses (MAD)
MeSH Terms: conditions — Hepatitis C | interventions — dasabuvir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1. ABT-333 Tablet (Active Comparator): Three 400mg ABT-333 Tablets, BID
  Interventions: Drug: ABT-333
- 2. ABT-333 Tablet (Active Comparator): Four 400mg ABT-333 Tablets, BID
  Interventions: Drug: ABT-333
- 3. Placebo (Placebo Comparator): Three or four placebo tablets, BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABT-333 — See arm description for more information
  Arms: 1. ABT-333 Tablet; 2. ABT-333 Tablet
Drug: Placebo — See arm description for more information
  Arms: 3. Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics of escalating multiple doses of the ABT-333 tablet formulation in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* overall healthy subjects between the ages of 18 to 55 years old;
* if female, subject must be either postmenopausal for at least 2 years or surgically sterile;
* females must have negative results for pregnancy tests performed;
* if male, subject must be surgically sterile or practicing at least 1 of the following methods of birth control:

  * partner(s) using IUD,
  * partner(s) using oral, injected or implanted methods of hormonal contraceptives,
  * subject and/or partner(s) using double-barrier method;
* Body Mass Index is 18 to 29, inclusive

Exclusion Criteria:

* history of significant sensitivity to any drug;
* positive test for HAV IgM, HBsAg, HCV Ab or HIV Ab;
* history of gastrointestinal issues or procedures;
* history of seizures, diabetes or cancer (except basal cell carcinoma);
* clinically significant cardiovascular, respiratory (except mild asthma), renal, gastrointestinal, hematologic, neurologic, thyroid, or any uncontrolled medical illness or psychiatric disorder;
* use of tobacco or nicotine-containing products with the 6-month period prior to study drug administration;
* donation or loss of 550 mL or more blood volume or receipt of a transfusion of any blood product within 8 weeks prior to study drug administration;
* clinically significant abnormal screening laboratory analyses and ECGs:

  * ALT > ULN,
  * AST > ULN,
  * ECG with QTcF>450 msec in females and >430 msec in males,
  * or ECG with 2nd or 3rd degree atrioventricular block;
* current enrollment in another clinical study;
* previous enrollment in this study;
* recent (6-month) history of drug/alcohol abuse that could preclude adherence to the protocol;
* pregnant or breastfeeding female;
* requirement for any OTC and/or prescription medication, vitamins and/or herbal supplements on a regular basis or use within the 2-week period prior to the first dose of study drug administration or within 10 half-lives of the respective medication;
* use of known inhibitors or inducers of cytochrome P450 3A or cytochrome P450 2C8 within 1 month prior to study drug administration;
* positive screen for drugs of abuse, alcohol, or cotinine;
* receipt of any drug by injection within 30 days prior to study drug administration;
* receipt of any investigational product within a time period equal to 10 half-lives of the product or a minimum of 6 weeks prior to study drug administration;
* consumption of alcohol within 48 hours prior to study drug administration;
* consumption of grapefruit, grapefruit products, star fruit, or star fruit products within the 72-hour period prior to study drug administration;
* consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive ABT-333;
* history of cardiac disease, including family history of long-QT syndrome or unexplained sudden death.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-05; Primary Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To assess multiple dose safety and tolerability of an ABT-333 tablet formulation relative to placebo by the evaluation of vital signs, ECGs, physical exams, clinical lab testing and adverse event monitoring. | 10 days
Values for the pharmacokinetic parameters of ABT-333 will be evaluated after pre- and post-dose blood draws. | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cohen, MD, Study Director — Abbott
Locations (1):
- Site Reference ID/Investigator# 20081, Waukegan, Illinois, United States